CLINICAL TRIAL: NCT05194020
Title: All in Dads! Program Evaluation
Brief Title: All in Dads! Healthy Marriage and Responsible Fatherhood Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Action for Children (Unknown)
Responsible Party: Principal Investigator, Matt Shepherd, Principal Investigator, Midwest Evaluation & Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002/03/30
Record Dates: First submitted 2021-11-22; First posted 2022-01-18 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Fathers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Services (Experimental): Participants receive 16 hours of Father Factor curricula, 4 hours of The New Playbook curricula, 4 hours of Money Smart curricula over the course of five weeks. Participants also receive on-going job readiness support and post-employment support.
  Interventions: Other: Primary Services

INTERVENTIONS:
Other: Primary Services — Participants receive 16 hours of Father Factor curricula, 4 hours of The New Playbook curricula, 4 hours of Money Smart curricula over the course of five weeks. Participants also receive on-going job readiness support and post-employment support.

SUMMARY:
The purpose of this study is to help fathers establish and strengthen their relationship with their children and the mothers of their children; to reduce domestic violence in vulnerable families; to improve economic stability of fathers through comprehensive, job-driven career services; to employ intensive case management barrier removal, individual job coaching, and comprehensive family development to improve short and long-term outcomes.

DETAILED DESCRIPTION:
After being informed about the study and giving consent, participants will enroll in a five-week All in Dads! program that collects data at enrollment, at the end of the program, and 12 months following the program. Research questions in this study are framed by a Descriptive Evaluation Design to assess whether outcomes improve for low-income fathers who participate in the All in Dads! (AID!) Project. Primary and secondary outcomes are assessed before and after participants complete core curricula-Father Factor, The New Playbook, and Money Smart-and Job Readiness Coaching and Career Development as employment support services (pre to post). Primary outcome measures will indicate whether behavior improved for healthy family relationships (parent, co-parent, and partner) and economic stability (financial, employment). Secondary outcome measures will indicate whether behavior improved for the attitudes and expectations that facilitate and reflect behavior for healthy family relationships and economic stability.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and older)
* Father/father figure
* Reside in Franklin County, Ohio

Exclusion Criteria:

* Minor (under the age of 18)
* Not a father/father figure
* Reside outside of Franklin County, Ohio

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 731 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2025-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation & Research
Locations (1):
- Action for Children, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. The study looks at data as a whole.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Services
Started (This is the number of participants who enrolled into the program.) | 720
Baseline Survey Completion (This is the number of participants enrolled into the study who completed the baseline survey.) | 697
Post Program Survey Completion (This is the number of participants who completed the post-program survey. It was not required to take the baseline survey to complete the post-program survey.) | 504
12-Month Follow-Up Survey Completion (We still collected a follow-up survey from participants who did not complete the program if we were able to reach them. Participants were not required to have completed the post-program survey to take the follow-up, but needed to have taken the baseline survey.) | 532
Completed | 720
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline is number of participants who consented to be in the study.
Arm/Group | Primary Services
Number analyzed (Participants) | 720
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 718
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 36.30 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 720
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43
  Not Hispanic or Latino | 662
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 524
  White | 127
  More than one race | 57
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 720

OUTCOME MEASURES:

1. Primary Outcome: Healthy Parenting Behavior Measurement #1
Description: 1A) Will participants report significantly healthier parenting behavior after completing primary educational services and employment support services?
  7 items engage w/child measured on the Healthy Parenting Behavior Scale #1.
  The scale was 1-5 and as follows:
  1=Never, 2=1 to 2 days per month, 3=3 or 4 days per month, 4=2 or 3 days per week, 5=Every day or almost every day
  1 item- frequency reach out to children (categories, 4-point scale); Measured on the Healthy Parenting Behavior Scale #2
  1=Every day or almost every day, 2=One to three times a week, 3=One to three times in the past month, 4=Never in the past month
  The 8 items are measured as a construct. All items are added together and divided by 8 to create the construct score. The higher the score, the better the outcome.
  maximum score of 4.5, minimum score of 1.0
Time Frame: Change in mean from baseline in behavior in parenting behavior (interaction with children) to mean at 12 months from enrollment.
Population: 248 participants responded to at least 80% of the items in this measure.
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | Primary Services
Number analyzed (Participants) | 248
total score
  Mean at baseline | 3.96 (.87)
  Mean at follow-up | 4.12 (.87)

2. Primary Outcome: Healthy Co-parenting Behavior Measurement #1
Description: 2) Will participants report significantly healthier co-parenting behavior after completing primary educational services and employment support services?
  Co-parenting behavior:
  11 items: frequency of agreement with key co-parenting behaviors (interval, 5-point scale)
  Measured on the Healthy Co-Parenting Behavior Scale #1 as:
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  Individually, for five items, the higher the score the better. Six items are reverse scored, the lower the rating, the better the score.
  The construct is created by adding all scores together and dividing by 11. The higher the score on a scale of 1-5, the better the outcome. The lower the score, the worse the outcome.
Time Frame: Change from baseline in co-parenting behavior at 12 months from enrollment.
Population: 468 participants responded to at least 80% of the items in this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Services
Number analyzed (Participants) | 468
score on a scale
  Mean at Baseline | 3.30 (1.17)
  Mean at Follow-Up | 3.39 (1.07)

3. Primary Outcome: Healthy Financial Behavior Measurement #1
Description: 3) Will participants report significantly healthier financial behavior after completing primary educational services and employment support services?
  Father financial behavior:
  2 items: yes or no questions for have resume, checking/savings accounts (dichotomous)
  Numbers reported in the results are counts of yes (participant has a checking account and participant has a savings account).
Time Frame: Change from baseline in father financial behavior at 12 months from enrollment.
Population: 507 participants responded to at least 80% of the items in this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Services
Number analyzed (Participants) | 507
Participants
  Number of participants with checking account at baseline | 356
  Number of participants with checking account at 12-month follow-up | 432
  Number of participants with savings account at baseline | 278
  Number of participants with savings account at 12-month follow-up | 352

4. Secondary Outcome: Healthy Parenting Attitudes Measurement #1
Description: 4) Will participants report significantly healthier parenting attitudes after completing primary educational services and employment support services?
  Parenting attitudes (toward children) 7 items: frequency of key attitudes (categories, 5-point scale)
  Measured on the Healthy Parenting Attitudes Scale #1 as:
  1. Always
  2. Often
  3. Sometimes
  4. Rarely
  5. Never
  A construct is created by adding the score of the 7 items together and dividing by 7.
  Maximum score=5 (7*5/7), minimum score=1.0 (1*7/7)
Time Frame: Change in parenting attitudes (towards children) from enrollment to completion of the program (post-survey).
Population: 331 participants responded to at least 80% of the items in this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Services
Number analyzed (Participants) | 331
score on a scale
  Mean at Baseline | 4.56 (.44)
  Mean at Post-Program Survey | 4.59 (.41)

ADVERSE EVENTS:
Time Frame: 1 year through study completion
Description: The definitions of adverse events do not differ from the clinicaltrials.gov definitions.
Arm/Group | Primary Services
All-Cause Mortality (participants affected / at risk) | 0/720
Serious Adverse Events (participants affected / at risk) | 0/720
Other Adverse Events (participants affected / at risk) | 0/720

LIMITATIONS AND CAVEATS:
High levels of attrition due to items not being applicable to some participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT05194020/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT05194020/SAP_001.pdf